CLINICAL TRIAL: NCT03861481
Title: A Multicenter, Randomized, Subject-Blind, Investigator-Blind, Placebo-Controlled, Parallel-Group Study Evaluating the Efficacy, Safety, and Tolerability of Rozanolixizumab in Subjects With Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Brief Title: A Study to Assess the Efficacy, Safety and Tolerability of Rozanolixizumab in Subjects With Chronic Inflammatory Demyelinating Polyradiculoneuropathy
Acronym: MyCIDPchoice
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CIDP01; 2016-002411-17 (EudraCT Number)
Expanded Access: NCT05014724 (No longer available)
Record Dates: First submitted 2019-03-01; First posted 2019-03-04 (Actual); Results first posted 2022-04-04 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP)
Keywords: Chronic inflammatory demyelinating polyradiculoneuropathy; CIDP; UCB7665; rozanolixizumab
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — rozanolixizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Rozanolixizumab (Experimental): Subjects will be randomized to receive predefined subcutaneous doses of rozanolixizumab at a specified frequency
  Interventions: Drug: Rozanolixizumab
- Placebo (Placebo Comparator): Subjects will be randomized to receive predefined subcutaneous doses of placebo at a specified frequency
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rozanolixizumab — Subjects will receive rozanolixizumab in a specified sequence during the treatment period.
  Arms: Rozanolixizumab
Other: Placebo — Subjects will receive placebo in a specified sequence during the treatment period.
  Arms: Placebo

SUMMARY:
The purpose of the study is to evaluate clinical efficacy of rozanolixizumab as a treatment for subjects with chronic inflammatory demyelinating polyradiculoneuropathy (CIDP).

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥ 18 years of age with a minimum body weight of ≥42 kg at Visit 1 (Screening)
* Subject has a documented definite or probable diagnosis of Chronic Inflammatory Demyelinating Polyradiculoneuropathy (CIDP) according to the European Federation of Neurological Societies (EFNS)/ Peripheral Nerve Society (PNS) criteria 2010
* Subject has an immunoglobulin-dependency confirmed by clinical examination during therapy or upon interruption or reduction of therapy within 18 months prior to Screening and documented in medical history
* Subject is on a stable dosage (not more than ±20% deviation) for subcutaneous immunoglobulin (SCIg) or intravenous immunoglobulin (IVIg) and a fixed interval for at least 4 months of either treatment
* Female subjects of childbearing potential must agree to use a highly effective method of birth control, during the study and for a period of 3 months after their final dose of investigational medicinal product (IMP)
* Male subjects with a partner of childbearing potential must be willing to use a condom when sexually active during the study and for 3 months after the final administration of IMP

Exclusion Criteria:

* Previously received treatment in this study or subject has previously been exposed to rozanolixizumab
* Current diagnosis or has a history of Type 1 or Type 2 diabetes mellitus and/or hemoglobin A1c level >6.0 %
* Known immunoglobulin M (IgM)-mediated neuropathy
* Clinical or known evidence of associated systemic diseases that might cause neuropathy or treatment with agents that might lead to neuropathy
* History of clinically relevant ongoing chronic infections
* Family history of primary immunodeficiency
* Received a live vaccination within 8 weeks prior to the Baseline Visit; or intends to have a live vaccination during the course of the study or within 7 weeks following the final dose of IMP
* Received any experimental biological agent within or outside of a clinical study in the past 3 months or within 5 half-lives prior to Baseline
* Prior treatment with rituximab, ofatumumab, or ocrelizumab in the 6 months prior to the Baseline Visit or subject has had prior treatment with rituximab, ofatumumab, or ocrelizumab in the 12 months prior to Baseline and B cells are not within the normal range
* Female subject who is pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (22):
- United States (7):
  - Cidp01 902, Phoenix, Arizona
  - Cidp01 905, Los Angeles, California
  - Cidp01 901, Tampa, Florida
  - Cidp01 907, Augusta, Georgia
  - Cidp01 911, Lexington, Kentucky
  - Cidp01 903, Charlotte, North Carolina
  - Cidp01 912, Durham, North Carolina
- Belgium (3):
  - Cidp01 101, Ghent
  - Cidp01 102, Leuven
  - Cidp01 103, Liège
- Cidp01 302, Copenhagen, Denmark
- France (3):
  - Cidp01 402, Bordeaux
  - Cidp01 404, Nice
  - Cidp01 401, Strasbourg
- Germany (4):
  - Cidp01 501, Berlin
  - Cidp01 503, Essen
  - Cidp01 505, Göttingen
  - Cidp01 502, Würzburg
- Cidp01 601, Amsterdam, Netherlands
- Spain (2):
  - Cidp01 701, Barcelona
  - Cidp01 702, Barcelona
- Cidp01 802, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll study participants in March 2019 and concluded in March 2021.
Pre-assignment Details: Participant Flow refers to the Randomized Set.
Groups:
- Placebo: Participants received placebo matched to rozanolixizumab as a subcutaneous injection once weekly for 12 weeks.
- Rozanolixizumab: Participants received rozanolixizumab Dose A as a subcutaneous injection once weekly for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Rozanolixizumab
Started | 17 | 17
Completed | 11 | 10
Not Completed | 6 | 7
Not completed — COVID-19 pandemic circumstances | 0 | 1
Not completed — Participant not plan to participate in the study CIDP04 | 1 | 0
Not completed — Relapse | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lack of Efficacy | 4 | 5

BASELINE CHARACTERISTICS:
Population: The Randomized Set consisted of all participants randomized into the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Rozanolixizumab | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 12 | 28
  >=65 years | 1 | 5 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.4 (7.4) | 57.3 (13.3) | 56.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 9 | 9 | 18
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 0 | 1
  Black | 1 | 1 | 2
  White | 11 | 15 | 26
  Other/mixed | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 13 (Day 85) in Inflammatory Rasch-built Overall Disability Scale (iRODS) Score
Description: iRODS is a linearly weighted patient-reported outcome measure (questionnaire) that captures activity and social participation limitations in participants with chronic inflammatory demyelinating polyradiculoneuropathy. Questionnaire consisted of 24 items (including eating, taking a shower, walking a flight of stairs, standing for hours, etc.) and assesses a participant's ability to perform daily and social activities. Participants had 3 response options: 0=impossible to perform; 1=performed with difficulty; 2=easily performed, performed without difficulty. Raw sum scores of iRODS (range 0 to 48, where 0=worse and 48=best) were translated to log odds units (logits) scale, placing participant' estimates on same logit scale, which had a score range of -6.95 (most severe activity and social participation restrictions) to 8.11 (no activity and social participation limitations). A positive change is associated with a better outcome of less disease activity and more social activity.
Time Frame: From Baseline up to Week 13 (Day 85)
Population: The Full Analysis Set (FAS) consisted of all participants who received at least one dose of treatment and who had a Baseline and at least one valid post-Baseline iRODS measurement up to Week 13 (Day 85)/premature end of treatment (inclusively).
Measure: Least Squares Mean (Standard Error); unit: score on a scale (logits)
Arm/Group | Placebo | Rozanolixizumab
Number analyzed (Participants) | 17 | 16
score on a scale (logits) | 0.234 (0.379) | 0.181 (0.468)
Statistical Analysis 1: Comparison: Placebo vs Rozanolixizumab; Test type: Superiority; LS Mean difference (Rozimab - Placebo) = -0.052, 90% CI 2-sided [-0.892 to 0.788] — MMRM analysis (fixed effect terms: treatment, baseline iRODS score, prior Ig therapy administration route, assessment week, treatment by week interaction; random effect term: study participant). LS Mean Difference > 0 favours rozanolixizumab

ADVERSE EVENTS:
Time Frame: From Baseline until the Safety Follow-up Visit (up to Week 24)
Description: A TEAE is defined as any event that was not present prior the first administration of IMP or any unresolved event already present before the first administration of IMP that worsens in intensity following exposure to treatment until 8 weeks following the last administration of IMP.
Arm/Group | Placebo | Rozanolixizumab
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 2/17
Other Adverse Events (participants affected / at risk) | 14/17 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Rozanolixizumab (N=17)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=17) | Rozanolixizumab (N=17)
Diarrhoea (Gastrointestinal disorders) | 3 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (6) | 0 (0)
Infusion site erythema (General disorders) | 0 (0) | 3 (4)
Peripheral swelling (General disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 3 (3) | 0 (0)
Pain (General disorders) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Bacterial test positive (Investigations) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 5 (10) | 6 (9)
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 4 (4) | 4 (4)
Hypoaesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2019-07-09): https://cdn.clinicaltrials.gov/large-docs/81/NCT03861481/Prot_002.pdf
  • Statistical Analysis Plan (2021-04-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT03861481/SAP_001.pdf